CLINICAL TRIAL: NCT03730129
Title: A Prospective Case Series of Subcutaneous Immunoglobulin for Prophylaxis of Infections in Patients With Chronic Lymphocytic Leukemia With Impaired Humoral Immunity
Brief Title: Humoral Immunodeficiency in CLL and Therapy With Subcutaneous Ig
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, S. Shahzad Mustafa, Associate Medical Director, Rochester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIC1850-A-18
Record Dates: First submitted 2018-10-11; First posted 2018-11-05 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Secondary Immune Deficiency Disorder
Keywords: chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ig replacement (Experimental): Subjects will receive Hizentra 0.4 mg/kg subq once weekly.
  Interventions: Drug: Hizentra

INTERVENTIONS:
Drug: Hizentra — Subjects will receive Hizentra 0.4 mg/kg qweekly subcutaneously for 6 months (24 weeks)

SUMMARY:
Patients with chronic lymphocytic leukemia (CLL) are at increased risk of infections as compared to age matched controls, with infections being a major cause of morbidity and mortality. Previous studies have shown that patients with CLL have both hypogammaglobinemia and impaired humoral immunity as defined by vaccine responses to both polysaccharide and peptide antigens. Attempts at decreasing infections in CLL have included therapy with prophylactic antibiotics and intravenous immunoglobulin. In general clinical practice and in previous studies, patients have started IV immunoglobulin replacement therapy if they have a history of serious infection or hypogammaglobinemia (defined as Immunoglobulin G below 500-600 g/dL), but vaccine responses have not been evaluated. This study will identify CLL patients with humoral immunodeficiency by checking both Ig levels and vaccines responses. In patients with impaired humoral immunity, the investigators will use subcutaneous immunoglobulin replacement to show this intervention will increase Ig levels, protective antibody titers, and be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia
* Medically stable, with expected survival of > 1 year
* Able to understand and willingness to sign a written informed consent
* Able to comply with study procedures

Exclusion Criteria:

* Previously diagnosed primary immunodeficiency
* Additional immunosuppressive states as assessed by the primary or co investigators
* Ongoing therapy with Ig replacement
* Serum IgG < 500 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Identify patients with CLL with humoral immunodeficiency despite serum IgG > 500 mg/dL. | 10 months
  Incidence of humoral immunodeficiency
Number of patients who increase IgG to above 700 mg/dL | 10 months
  Effectiveness of Hizentra to change IgG levels

SECONDARY OUTCOMES:
Number of patients who increase diphtheria IgG to above 0.1 IU/mL, tetanus IgG to above 0.1 IU/mL, and IgG to streptococcus pneumonia to above 1.3 mcg/mL | 10 months
  Effectiveness of Hizentra to change specific antibody titers in CLL
Number of subjects with treatment-related adverse effects as assessed by CTCAE v4.0 | 10 months
  Safety and tolerability of Hizentra in CLL
Quality of life (Short Form 36) on subcutaneous Ig replacement therapy a 0-100 scale, with lower scores indicating higher disability/lower quality of life | 10 months
  Does Hizentra change quality of life scores in patients with CLL
Track the number of infections requiring antibiotics, further characterized per severity as defined in previous studies | 10 months
  Does Hizentra change the rate of non-neutropenic infections in CLL

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Mustafa, MD, Principal Investigator — Rochester General Hospital
Locations (1):
- Allergy, Immunology, Rheumatology at Rochester Regional Health, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twomey JJ. Infections complicating multiple myeloma and chronic lymphocytic leukemia. Arch Intern Med. 1973 Oct;132(4):562-5. No abstract available. PMID 4542660
- [Background] Oscier D, Dearden C, Eren E, Fegan C, Follows G, Hillmen P, Illidge T, Matutes E, Milligan DW, Pettitt A, Schuh A, Wimperis J; British Committee for Standards in Haematology. Guidelines on the diagnosis, investigation and management of chronic lymphocytic leukaemia. Br J Haematol. 2012 Dec;159(5):541-64. doi: 10.1111/bjh.12067. Epub 2012 Oct 11. No abstract available. PMID 23057493
- [Background] Lachance S, Christofides AL, Lee JK, Sehn LH, Ritchie BC, Shustik C, Stewart DA, Toze CL, Haddad E, Vinh DC. A Canadian perspective on the use of immunoglobulin therapy to reduce infectious complications in chronic lymphocytic leukemia. Curr Oncol. 2016 Feb;23(1):42-51. doi: 10.3747/co.23.2810. Epub 2016 Feb 18. PMID 26966403
- [Background] Chapel H, Dicato M, Gamm H, Brennan V, Ries F, Bunch C, Lee M. Immunoglobulin replacement in patients with chronic lymphocytic leukaemia: a comparison of two dose regimes. Br J Haematol. 1994 Sep;88(1):209-12. doi: 10.1111/j.1365-2141.1994.tb05002.x. PMID 7803248
- [Background] Dicato M, Chapel H, Gamm H, Lee M, Ries F, Marichal S, Wirth C, Griffith H, Brennan V. Use of intravenous immunoglobulin in chronic lymphocytic leukemia. A brief review. Cancer. 1991 Sep 15;68(6 Suppl):1437-9. doi: 10.1002/1097-0142(19910915)68:6+3.0.co;2-h. PMID 1878842
- [Background] Molica S, Musto P, Chiurazzi F, Specchia G, Brugiatelli M, Cicoira L, Levato D, Nobile F, Carotenuto M, Liso V, Rotoli B. Prophylaxis against infections with low-dose intravenous immunoglobulins (IVIG) in chronic lymphocytic leukemia. Results of a crossover study. Haematologica. 1996 Mar-Apr;81(2):121-6. PMID 8641639
- [Background] Raanani P, Gafter-Gvili A, Paul M, Ben-Bassat I, Leibovici L, Shpilberg O. Immunoglobulin prophylaxis in hematological malignancies and hematopoietic stem cell transplantation. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD006501. doi: 10.1002/14651858.CD006501.pub2. PMID 18843719
- [Background] Dhalla F, Lucas M, Schuh A, Bhole M, Jain R, Patel SY, Misbah S, Chapel H. Antibody deficiency secondary to chronic lymphocytic leukemia: Should patients be treated with prophylactic replacement immunoglobulin? J Clin Immunol. 2014 Apr;34(3):277-82. doi: 10.1007/s10875-014-9995-5. Epub 2014 Feb 21. PMID 24557494
- [Background] Ueda M, Berger M, Gale RP, Lazarus HM. Immunoglobulin therapy in hematologic neoplasms and after hematopoietic cell transplantation. Blood Rev. 2018 Mar;32(2):106-115. doi: 10.1016/j.blre.2017.09.003. Epub 2017 Sep 19. PMID 28958644
- [Background] Sanchez-Ramon S, Dhalla F, Chapel H. Challenges in the Role of Gammaglobulin Replacement Therapy and Vaccination Strategies for Hematological Malignancy. Front Immunol. 2016 Aug 22;7:317. doi: 10.3389/fimmu.2016.00317. eCollection 2016. PMID 27597852
- [Background] Friman V, Winqvist O, Blimark C, Langerbeins P, Chapel H, Dhalla F. Secondary immunodeficiency in lymphoproliferative malignancies. Hematol Oncol. 2016 Sep;34(3):121-32. doi: 10.1002/hon.2323. Epub 2016 Jul 12. PMID 27402426
- [Background] Cooperative Group for the Study of Immunoglobulin in Chronic Lymphocytic Leukemia; Gale RP, Chapel HM, Bunch C, Rai KR, Foon K, Courter SG, Tait D. Intravenous immunoglobulin for the prevention of infection in chronic lymphocytic leukemia. A randomized, controlled clinical trial. N Engl J Med. 1988 Oct 6;319(14):902-7. doi: 10.1056/NEJM198810063191403. PMID 2901668
- [Background] Looney RJ, Huggins J. Use of intravenous immunoglobulin G (IVIG). Best Pract Res Clin Haematol. 2006;19(1):3-25. doi: 10.1016/j.beha.2005.01.032. PMID 16377538
- [Background] Berger M. Adverse effects of IgG therapy. J Allergy Clin Immunol Pract. 2013 Nov-Dec;1(6):558-66. doi: 10.1016/j.jaip.2013.09.012. Epub 2013 Oct 31. PMID 24565701
- [Background] Gardulf A. Immunoglobulin treatment for primary antibody deficiencies: advantages of the subcutaneous route. BioDrugs. 2007;21(2):105-16. doi: 10.2165/00063030-200721020-00005. PMID 17402794
- [Background] Lingman-Framme J, Fasth A. Subcutaneous immunoglobulin for primary and secondary immunodeficiencies: an evidence-based review. Drugs. 2013 Aug;73(12):1307-19. doi: 10.1007/s40265-013-0094-3. PMID 23861187
- [Background] Compagno N, Cinetto F, Semenzato G, Agostini C. Subcutaneous immunoglobulin in lymphoproliferative disorders and rituximab-related secondary hypogammaglobulinemia: a single-center experience in 61 patients. Haematologica. 2014 Jun;99(6):1101-6. doi: 10.3324/haematol.2013.101261. Epub 2014 Mar 28. PMID 24682509
- [Background] Vacca A, Melaccio A, Sportelli A, Solimando AG, Dammacco F, Ria R. Subcutaneous immunoglobulins in patients with multiple myeloma and secondary hypogammaglobulinemia: a randomized trial. Clin Immunol. 2018 Jun;191:110-115. doi: 10.1016/j.clim.2017.11.014. Epub 2017 Nov 28. PMID 29191714
- [Derived] Mustafa SS, Jamshed S, Vadamalai K, Ramsey A. Subcutaneous immunoglobulin replacement for treatment of humoral immune dysfunction in patients with chronic lymphocytic leukemia. PLoS One. 2021 Oct 15;16(10):e0258529. doi: 10.1371/journal.pone.0258529. eCollection 2021. PMID 34653210